CLINICAL TRIAL: NCT06811285
Title: The Effect of Kinesiological Taping and Foot Massage Applied to Postpartum Women After Cesarean Delivery on Pain, Fatigue, and Mood: A Randomized Controlled Trial
Brief Title: Kinesio Taping and Foot Massage for Post-Cesarean Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Kevser Gürsan, Dr., Uşak University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 477-477-24
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Pain; Fatigue; Mood (Psychological Function); Postpartum Women
Keywords: Pain; Fatigue; Mood; Postpartum women
MeSH Terms: conditions — Pain; Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinesiological Taping Group (Experimental): The Kinesiological Taping group will receive two parallel I-shaped kinesiological taping applications.
  Interventions: Other: Kinesiological Taping
- Foot Massage Group (Experimental): The Foot Massage Group will receive foot massage for 20 minutes.
- Control Group (No Intervention): No intervention will be applied.

INTERVENTIONS:
Other: Kinesiological Taping — The Kinesiological Taping group will receive two parallel I-shaped kinesiological taping applications.
  Arms: Kinesiological Taping Group
Other: Foot Massage Group — The Foot Massage Group will receive foot massage for 20 minutes.

SUMMARY:
After a cesarean section, postpartum women may experience pain, fatigue, and various negative mood disturbances. These effects pose a significant public health concern by threatening both maternal and infant health. To prevent these public health problems, it is essential to improve maternal health and well-being. This randomized controlled trial aims to conduct a comparative investigation into the effects of kinesiological taping and foot massage on postpartum pain, fatigue, and mood in women who have undergone cesarean delivery.

The primary research questions are as follows:

Does the application of kinesiological taping to postpartum women after cesarean section influence pain, fatigue, and mood? Does the application of foot massage to postpartum women after cesarean section influence pain, fatigue, and mood? To address these questions, the study will involve postpartum women who meet the inclusion criteria and provide informed consent. Participants will be randomly assigned to three groups: one group will receive kinesiological taping, another will receive foot massage, and the control group will not receive any intervention. In postpartum women, pain levels will be assessed at postoperative hours 8, 9, 33, and 34. Fatigue and mood will be evaluated at postoperative hour 8 (prior to the intervention) and hour 34.

DETAILED DESCRIPTION:
Cesarean delivery has become an increasingly common surgical method of birth among mothers in recent times. Over the years, global cesarean delivery rates have risen significantly. The significant increase in cesarean rates has highlighted the need for treatments aimed at alleviating pain complaints in postpartum women. Opioids and local anesthetics are frequently used in the treatment of these pain complaints. However, the use of these medications is often associated with side effects such as nausea, vomiting, itching, sedation, respiratory issues, and depression in mothers. To reduce or eliminate the side effects of these medications, there is a need for simple, practical, and non-pharmacological treatment approaches that can be implemented clinically.

In addition to the pain experienced after cesarean surgery, fatigue, the burden of caring for their newborns or themselves, hormonal changes, and other factors can contribute to various negative emotional effects in mothers. These issues pose a significant public health problem by threatening both maternal and neonatal health. Addressing these public health concerns is crucial to improving maternal health and well-being. In this regard, our study aims to investigate the effects of kinesiology taping and foot massage on pain, fatigue, and mood in mothers following cesarean delivery through a randomized controlled trial. In the study, some mothers who have undergone cesarean delivery will receive kinesiology taping, others will undergo foot massage, and the remaining group will receive no intervention.

Kinesiology taping is one of the non-pharmacological methods that has gained increasing use across various disciplines for pain management. It is a therapeutic technique based on the body's natural healing process. The technique is applied according to Kase's principles, and as a result, fascial tissue healing occurs, pain and edema are reduced, and tissue blood circulation is enhanced. Foot massage, when applied to mothers after cesarean delivery, may help reduce pain and fatigue, thus promoting a general sense of well-being. The mechanism of foot massage involves stimulating the nociceptors beneath the skin of the foot, which may be effective in pain reduction. Based on this, we aim to compare the effects of kinesiology taping and foot massage on pain, fatigue, and mood in post-cesarean mothers.

The study group will consist of mothers who have undergone cesarean delivery, meet the research criteria, and have agreed to participate in the study after receiving detailed information. Participants will complete an introductory information form, and their pain will be assessed using the Visual Analog Scale, fatigue will be assessed using the Visual Analog Scale for Fatigue (VAS-F), and mood will be assessed using the Brief Mood Introspection Scale (BMIS). Before starting the intervention, the study group will be randomly divided into three groups. Randomization will be performed using www.randomizer.org. One group will receive kinesiology taping, another will receive foot massage, and the control group will receive no intervention. Pain, fatigue, and mood assessments will be performed before any intervention at post-operative hour 8. Pain assessments will be conducted at post-operative hour 9, post-operative hour 33, and post-operative hour 34 for all groups. Fatigue and mood assessments will be made at post-operative hour 34.

For the kinesiology taping group, the taping will be applied bilaterally in a parallel "I" shape on the rectus abdominis muscles. Pain measurements will be taken one hour after the application (post-op hour 9), at 24 hours (post-op hour 33), and after the tape is removed (post-op hour 34). The effect of kinesiology taping on pain will also be assessed at post-op hour 33.

For the foot massage intervention, each foot will receive manual massage for 10 minutes, totaling 20 minutes, with two applications in total. The first foot massage will be administered at post-op hour 9, and immediate pain measurements will be taken. The second foot massage will be applied at post-op hour 33, followed by immediate pain measurements and one-hour follow-up measurements at post-op hour 34. The control group will only have pain assessments at post-op hours 8, 9, 33, and 34. The data obtained from these evaluations will undergo statistical analysis to determine which intervention is more effective for each variable.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 18-45,
* Being able to speak Turkish and to express oneself in Turkish,
* Having undergone a pregnancy duration of 38-42 weeks,
* Have given birth via cesarean section,
* Have undergone a transverse incision,
* To give live birth, delivered a baby weighing between 2500 and 4000 grams,
* Having a singleton pregnancy,
* The analgesics used should be of the same type and administered in the same dose,
* Not having dermatological issues.
* No mental disability or perception problems,
* No communication difficulties,
* Be willing to participate in the study.

Exclusion Criteria:

* Having been diagnosed with allergic skin conditions and developing postpartum complications (such as bleeding, infection, etc.),
* A body mass index of 40 or higher,
* Hemoglobin levels lower than 9 g/dL
* Hematocrit levels lower than 30%,
* Postpartum women who have experienced a neonatal anomaly,
* Women who have been diagnosed with any psychiatric disorder,
* Used different types and doses of analgesics in the postoperative period,
* Postpartum women whose infants are receiving treatment in the neonatal intensive care unit

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Postpartum women
Enrollment: 97 (Actual)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
Pain assessment | Between the 8th and 34th postoperative hours.
  In the study, the Visual Analog Scale (VAS) will be utilized to assess pain levels in postpartum women who have undergone a cesarean section. The VAS was developed by Price et al. in 1983 to evaluate subjective pain and has been widely accepted in the global literature as a reliable and easy-to-administer scale. The VAS consists of a 10 cm vertical or horizontal line with two endpoints labeled differently (0 = No pain at all - Completely comfortable, and 10 = Worst imaginable pain).

SECONDARY OUTCOMES:
Fatigue and energy assessment | Between the 8th and 34th postoperative hours.
  The Visual Analogue Scale for Fatigue (VAS-F) will be used to assess fatigue in postpartum women. VAS-F is used to measure energy and fatigue levels. It was developed by Lee et al. (1991) and consists of two subscales: fatigue (items 1, 2, 3, 4, 5, 11, 12, 13, 14, 15, 16, 17, and 18) and energy (items 6, 7, 8, 9, and 10), comprising a total of 18 items. The scale has been validated for assessing fatigue during pregnancy and the postpartum period in research settings. Each item is presented on a 10 cm horizontal line, with one end representing a positive statement and the other end representing a negative statement. In the fatigue subscale, items are arranged from positive to negative, whereas in the energy subscale, the order is reversed. The total score for the fatigue subscale ranges from 0 to 130, while the energy subscale scores range from 0 to 50. A higher score in the fatigue subscale and a lower score in the energy subscale indicate increased fatigue severity.
Mood assessment (Positive and negative ) | Between the 8th and 34th postoperative hours.
  The Brief Mood Introspection Scale (BMIS) was developed by Mayer and Gaschke in 1988 to assess participants' current mood states. This 16-item scale aims to evaluate both positive and negative mood levels. The positive mood subscale consists of eight items: cheerful, happy, compassionate, content, energetic, calm, loving, and active. Conversely, the negative mood subscale includes eight items: sad, fatigued, gloomy, tense, drowsy, irritable, nervous, and weary. The BMIS is a four-point Likert-type scale, where each item is rated from "definitely feel" (4 points) to "definitely do not feel" (1 point). Higher scores on either subscale indicate a higher intensity of positive or negative mood. The total possible score for each subscale ranges from a minimum of 8 to a maximum of 32.

CONTACTS AND LOCATIONS:
Overall Officials: Kevser Gursan, Dr, Principal Investigator — Uşak University
Locations (1):
- Usak University, Uşak, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No